CLINICAL TRIAL: NCT06776965
Title: Impact of Ultra-processed Foods in a Population of Patients With Chronic Rheumatic Diseases (Rheumatoid Arthritis, Spondyloarthritis, Osteoarthritis).
Brief Title: Ultra Processed Foods Consumption and Impact in Rheumatic Diseases.
Acronym: NUTRIRIC
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL24_0947; 2024-A02327-40 (Other: ID-RCB)
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Rheumatoid Arthritis; Spondyloarthritis; Osteoarthritis
Keywords: Ultra-processed food; osteoarthritis; rheumatoid arthritis; spondyloarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylarthritis; Osteoarthritis | interventions — Extravehicular Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Rheumatoid Arthritis: Patients in the first group will correspond to those with rheumatoid arthritis according to ACR criteria of RA
  Interventions: Other: Dietary Questionnaire; Other: Evaluation of disease activity (DAS-28, ASDAS, EVA, number of swollen joints, number of painful joint, nocturnal pain, morning stiffness)
- Spondyloarthritis: Patients in the second group will correspond to those with spondyloarthritis according ASDAS criteria
  Interventions: Other: Dietary Questionnaire; Other: Evaluation of disease activity (DAS-28, ASDAS, EVA, number of swollen joints, number of painful joint, nocturnal pain, morning stiffness)
- Osteoarthritis: Patients in the third group will correspond to those with spondyloarthritis according ACR criteria
  Interventions: Other: Dietary Questionnaire; Other: Evaluation of disease activity (DAS-28, ASDAS, EVA, number of swollen joints, number of painful joint, nocturnal pain, morning stiffness)
- Controls: Patients without rheumatic disease
  Interventions: Other: Dietary Questionnaire; Other: Evaluation of disease activity (DAS-28, ASDAS, EVA, number of swollen joints, number of painful joint, nocturnal pain, morning stiffness)

INTERVENTIONS:
Other: Dietary Questionnaire — Self administered dietary questionnaire at baseline, 6 and 12 months.
Other: Evaluation of disease activity (DAS-28, ASDAS, EVA, number of swollen joints, number of painful joint, nocturnal pain, morning stiffness) — Self administered questionnaire of disease activity at baseline, 6 and 12 months.

SUMMARY:
Ultra-processed foods (UPF) represent one of the mainstays of today's diet. They are defined by the NOVA classification system. It was demonstrated that UPF consumption was associated with activity of inflammatory bowel diseases with underlying mechanisms not fully identified yet. It is suspected that UPF constituents could modify the gut microbiota, increase intestinal barrier permeability and directly engage immune surveillance systems, effects that could individually or synergistically increase the risk of immunomediated diseases. As some pathophysiological mechanisms are shared among IBD and rheumatic diseases, we have wondered if UPF consumption could be associated with increased risk of rheumatic disease and/or with their activity.

Our primary aim will be to study the pattern of UPF consumption in patients with rheumatic diseases. Our secondary objectives will be to study the activity of diseases according to UPF consumption.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* chronic rheumatic disease (Rheumatoid arthritis, spondyloarthritis, osteoarthritis)
* ability to perform questionnaires

Exclusion Criteria:

* Judicial protection measure
* Refusal to participate in the study
* Suffering from 2 rheumatic disease simultaneously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic rheumatological diseases (spondylitis, rheumatoid arthritis, osteoarthritis) and control population (also followed for any other pathology in the department).
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Describe the consumption of ultra-processed foods in patients with chronic inflammatory rheumatism | At baseline
  Describes the consumption of ultra-processed foods in patients with chronic inflammatory rheumatism using a self-assessment questionnaire (Score UPF Nova Screener) completed at baseline, 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Maxime AUROUX, MD, Principal Investigator — Hôpital Edouard Herriot
Locations (1):
- Edouard Herriot Hospital, Lyon, France